CLINICAL TRIAL: NCT03363256
Title: Web-based Addiction Treatment: Cultural Adaptation With American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee Campbell, Associate Professor of Clinical Psychiatric Social Work, New York State Psychiatric Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7555; R34DA040831 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Substance Use Disorders
Keywords: Digital therapeutics; Adaptation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU+TES-NAV (Experimental): Standard outpatient addiction treatment plus Therapeutic Education System adapted for AI/AN
  Interventions: Behavioral: TES-NAV; Behavioral: TAU
- TAU (Active Comparator): Standard outpatient addiction treatment
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TES-NAV — Internet-delivered psychosocial treatment grounded in the community reinforcement approach plus contingency management adapted for AI/AN
  Arms: TAU+TES-NAV
Behavioral: TAU — Standard outpatient addiction treatment

SUMMARY:
The purpose of the current study is to evaluate the preliminary efficacy of the Therapeutic Education System-Native Version (TES-NAV) (an efficacious web-delivered psychosocial intervention for substance use disorders adapted with American Indians/Alaska Natives [AI/AN]) to determine whether a future large-scale effectiveness trial is warranted. Specifically, a randomized controlled trial among urban AI/AN (N=80) attending outpatient addiction treatment services will be conducted to (1) estimate preliminary effect size of 12 weeks of TES-NAV on substance use disorder outcomes; (2) explore relevant moderators of TES-NAV outcomes; and (3) assess cultural factors that may correspond to variation in outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Identify as American Indian or Alaska Native
* Recent alcohol or drug use
* Within first 30 days of current outpatient treatment episode

Exclusion Criteria:

* Planned treatment episode of less than 3 months
* Insufficient ability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Consecutive weeks of drug/alcohol abstinence | 12 weeks
  Number of consecutive weeks of abstinence from drugs and alcohol

CONTACTS AND LOCATIONS:
Locations (1):
- Native American Rehabilitation Association of the Northwest, Inc., Portland, Oregon, United States

REFERENCES:
- [Background] Campbell AN, Turrigiano E, Moore M, Miele GM, Rieckmann T, Hu MC, Kropp F, Ringor-Carty R, Nunes EV. Acceptability of a web-based community reinforcement approach for substance use disorders with treatment-seeking American Indians/Alaska Natives. Community Ment Health J. 2015 May;51(4):393-403. doi: 10.1007/s10597-014-9764-1. Epub 2014 Jul 15. PMID 25022913
- [Background] Campbell AN, Nunes EV, Matthews AG, Stitzer M, Miele GM, Polsky D, Turrigiano E, Walters S, McClure EA, Kyle TL, Wahle A, Van Veldhuisen P, Goldman B, Babcock D, Stabile PQ, Winhusen T, Ghitza UE. Internet-delivered treatment for substance abuse: a multisite randomized controlled trial. Am J Psychiatry. 2014 Jun;171(6):683-90. doi: 10.1176/appi.ajp.2014.13081055. PMID 24700332
- [Derived] Campbell ANC, Rieckmann T, Pavlicova M, Choo TH, Molina K, McDonell M, West AE, Daw R, Marsch LA, Venner KL. Culturally tailored digital therapeutic for substance use disorders with urban Indigenous people in the United States: A randomized controlled study. J Subst Use Addict Treat. 2023 Dec;155:209159. doi: 10.1016/j.josat.2023.209159. Epub 2023 Sep 9. PMID 37690525